CLINICAL TRIAL: NCT02750215
Title: A Phase 2 Study of Capmatinib (INC280) in NSCLC Patients With MET Exon 14 Alterations Who Have Received Prior MET Inhibitor
Brief Title: A Study of Capmatinib (INC280) in NSCLC Patients With MET Exon 14 Alterations Who Have Received Prior MET Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Rebecca Suk Heist, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-019
Record Dates: First submitted 2016-04-19; First posted 2016-04-25 (Estimated); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Malignant Non-small Cell Neoplasm of Lung Stage IV
Keywords: MET exon 14 skipping; Stage IV non-small cell lung cancer NSCLC
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capmatinib (INC280) (Experimental): Patients who fulfill eligibility criteria will be entered into the trial to receive capmatinib.
  After the screening procedures confirm participation in the research study. Participants will receive capmatinib PO BID, 21-day cycles
  Interventions: Drug: Capmatinib (INC280)

INTERVENTIONS:
Drug: Capmatinib (INC280) — treatment with Capmatinib (INC280)

SUMMARY:
This research study is studying capmatinib as a treatment for advanced non-small cell lung cancer with MET exon 14 skipping, where the participant has already received prior therapy with a MET inhibitor.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Capmatinib as a treatment for any disease.

In this research study, the investigators are using the study drug called Capmatinib. Capmatinib is a specific blocker of the cMET protein. This protein acts as a trigger to start a series of events in your cells in what is known as the C-Met pathway. Patients with MET exon 14 skipping have activation of the MET pathway. By blocking MET, Capmatinib may slow or stop the growth and/or survival of cancer cells. Capmatinib is not yet FDA approved for the treatment of people with this type of cancer. It is not known if capmatinib will be effective in people who have previously had other drugs that block the cMET pathway. This study will help us understand how capmatinib works in the body and what capmatinib does to cancer. Any potential harmful effects of capmatinib will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures.
* Age ≥ 18 years
* Histologically or cytologically confirmed non-small cell lung cancer, advanced, recurrent, or metastatic
* MET exon 14 skipping alteration by molecular testing (local testing is accepted for eligibility; all patients will have confirmation by NGS-rearrangement assay at MGH but this result is not necessary for eligibility; local molecular pathology result will suffice). This testing can be from any archival or fresh sample.
* Must have received prior platinum containing chemotherapy for advanced/metastatic non-small cell lung cancer, or have refused or be ineligible for such therapy. Prior neoadjuvant/adjuvant platinum containing chemotherapy will count has having received prior platinum, provided that disease recurred within 6 months of completion of neoadjuvant/adjuvant therapy.
* EGFR and ALK status must be known in all patients with adenocarcinoma histology. Patients with activating EGFR mutations or ALK translocations are excluded from this study, unless disease has progressed on all available, approved therapies targeting these alterations.
* At least one measurable lesion as defined by RECIST 1.1. A previously irradiated site lesion may only be counted as a target lesion if there is clear sign of progression since the irradiation.
* Must have received prior MET inhibitor as their immediately preceding therapy. There are no limits to the number of lines of prior therapy as long as prior MET inhibitor is the most recent therapy.
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03). Patients with any grade of alopecia are allowed to enter the study.
* Patients must have adequate organ function including the following laboratory values at the screening visit:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support
  * Platelets ≥ 75 x 109/L
  * Hemoglobin (Hgb) > 9 g/dL
  * Calculated creatinine clearance (using Cockcroft-Gault formula) > 45 mL/min
  * Total bilirubin ≤ 1.5 x ULN, except for patients with Gilbert's syndrome, who may only be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
  * Aspartate transaminase (AST) ≤ 3 x ULN, except for patients with liver metastasis, who are included if AST ≤ 5 x ULN
  * Alanine transaminase (ALT) ≤ 3 x ULN, except for patients with liver metastasis, who are only included if ALT ≤ 5 x ULN
  * Alkaline phosphatase (ALP) ≤ 5.0 x ULN
  * Asymptomatic serum amylase ≤ grade 2. Patients with grade 1 or grade 2 serum amylase at the beginning of the study must be confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
  * Serum lipase ≤ ULN
  * Patients must have the following laboratory values within the laboratory normal limits or corrected to within normal limits with supplements during screening:

    * Potassium
    * Magnesium
    * Phosphorus
    * Total calcium (corrected for serum albumin)
* ECOG performance status (PS) of 0 or 1
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

* Patients with known hypersensitivity to any of the excipients of INC280 (crospovidone, mannitol, microcrystalline cellulose, povidone, sodium lauryl sulfate, magnesium stearate, colloidal silicon dioxide, and various coating premixes).
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
* Presence or history of carcinomatous meningitis
* Presence or history of a malignant disease other than disease to be treated in current protocol that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, indolent malignancies that currently do not require treatment, and completely resected carcinoma in situ of any type
* Clinically significant, uncontrolled heart diseases.

  * Unstable angina within 6 months prior to screening
  * Myocardial infarction within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication (s) is allowed prior to screening
  * Ventricular arrhythmias
  * Supraventricular and nodal arrhythmias not controlled with medication
  * Other cardiac arrhythmia not controlled with medication
  * QTcF > 480 msec
* Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting INC280 or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting INC280 or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting INC280 is allowed
* Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting INC280 or who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the study ≥ 1 week after the procedure
* Patients receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with INC280 and for the duration of the study:

  * Strong and moderate inhibitors of CYP3A4
  * Strong inducers of CYP3A4
  * Proton pump inhibitors (PPI)
* Impairment of GI function or GI disease that may significantly alter the absorption of INC280 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
* Unable or unwilling to swallow tablets as per dosing schedule
* Patients receiving unstable or increasing doses of corticosteroids. If patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms other than CNS related, dose must have been stabilized (or decreasing) for at least 5 days before first dose of INC280
* Patients receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least 1 week before first dose of INC280, and for the duration of the study. Patients on non-enzyme-inducing anticonvulsants are eligible
* Previous anti-cancer and investigational agents within 4 weeks or ≤ 5 x half-life of the agent (whichever is longer) before first dose of INC280. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 4 weeks before first dose of INC280
* Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities that in the opinion of the investigator may increase the risk associated with study participation, or that may interfere with the interpretation of study results
* Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
* Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 7 days after stopping treatment. Highly effective contraception methods include:
* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject
* Combination of any two of the following (a+b or a+c, or b+c):

  * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate ≤ 1%), for example hormone vaginal ring or transdermal hormone contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking drug and for 7 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S. Heist, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Capmatinib (INC280): Patients who fulfill eligibility criteria will be entered into the trial to receive capmatinib.
  After the screening procedures confirm participation in the research study. Participants will receive capmatinib PO BID, 21-day cycles
  Capmatinib (INC280): treatment with Capmatinib (INC280)
Period: Overall Study
Arm/Group | Capmatinib (INC280)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years]
  Age | 70 [57 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Smoking History [Number; unit: participants]
  Never | 8
  Former | 11
  Current | 1
Tumor Histology [Number; unit: participants]
  Adenocarcinoma | 16
  Squamous | 2
  Sarcomatoid or poorly differentiated carcinoma | 2
MET alteration [Number; unit: participants]
  Amplification | 5
  Exon 14 skipping | 15
Previous Chemotherapy [Number; unit: participants]
  Yes | 11
  No | 9
Previous Immunotherapy [Number; unit: participants]
  Yes | 7
  No | 13
Number of previous lines of therapy [Number; unit: participants]
  1 | 9
  2 | 3
  3 or more | 8
Number of previous MET-targeted therapies [Number; unit: participants]
  1 | 17
  2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is a greater than or equal to 30% decrease in the sum of the longest diameter of target lesions. ORR = CR + PR.
Time Frame: through study completion, an average of 14 months
Measure: Number; unit: percentage of participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
percentage of participants | 10

2. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: through study completion, an average of 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
months | 5.5 [1.3 to 11.0]

3. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) will be defined as the percentage of participants with complete response, partial response, and stable disease at 12 weeks by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. Complete Response (CR) is the disappearance of all target lesions. Partial Response (PR) is a greater than or equal to 30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease, taking as reference the smallest sum diameters while on study. Progressive Disease (PD) is a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. DCR = CR + PR + SD.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
percentage of participants | 80

4. Secondary Outcome: Intracranial Response Rate
Description: Intracranial response rate (IRR) will be calculated based on response assessments in the brain for patients with measurable CNS disease at baseline by RECIST v 1.1 criteria. IRR is defined as the percentage of patients with a confirmed intracranial complete response (CR) or partial response (CR) at week 12. CR is the disappearance of all target lesions and PR is a greater than or equal to 30% decrease in the sum of the longest diameter of target lesions. IRR = CR + PR.
Time Frame: 12 weeks
Population: Only 4 out of 20 participants had measurable brain metastases.
Measure: Number; unit: percentage of participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 4
percentage of participants | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) will be calculated from the time of first assessment of complete response (CR) or partial response (PR) per RECIST 1.1 until the first occurrence of progressive disease (PD) or death. CR is the disappearance of all target lesions. PR is a greater than or equal to 30% decrease in the sum of the longest diameter of target lesions. PD is a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 6 months
Population: Only 2 of 22 participants had complete response (CR) or partial response (PR) per RECIST 1.1, thus they were the only ones analyzed for DOR.
Measure: Mean (Full Range); unit: months
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 2
months | 3.8 [2.0 to 5.5]

6. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive. OS time for patients who are alive at the end of the study or are lost to follow up will be censored at the time of last contact. OS will be estimated using the Kaplan-Meier method.
Time Frame: From date of registration through study completion, an average of 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
months | 11.3 [5.5 to NA] — Upper limit was not reached due to an insufficient number of participants with events.

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events by Grade
Time Frame: From date of treatment start through study completion, an average of 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Participants
  Grade 3 | 8
  Grade 4 | 0
  Grade 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the treatment start date through study completion, an average of 14 months
Arm/Group | Capmatinib (INC280)
All-Cause Mortality (participants affected / at risk) | 15/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib (INC280) (N=20)
Hip fracture (Injury, poisoning and procedural complications) | 1
Edema limbs (General disorders) | 1
Wound infection (Injury, poisoning and procedural complications) | 1 — surgical wound infection
seizure (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1 — ischemic stroke
Thromboembolic event (Vascular disorders) | 1 — pulmonary embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib (INC280) (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Serum amylase increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 3
Atrioventricular block first degree (Cardiac disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 4
Diarrhea (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Reproductive system and breast disorders) | 1
Fatigue (General disorders) | 7
Blood bilirubin increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Lipase increased (Investigations) | 4
Edema limbs (General disorders) | 13
myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Platelet count decreased (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight gain (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT02750215/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT02750215/ICF_001.pdf